CLINICAL TRIAL: NCT00441753
Title: Cerebral Bloodflow and Carbondioxide Reactivity During Mild Therapeutic Hypothermia in Patients After Cardiac Arrest
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Radboud UNiversity Nijmegen Medical Centre, Radboud UNiversity Nijmegen Medical Centre
Other Study IDs: KSCH0601
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Cardiac Arrest; Post-Anoxic Encephalopathy
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Survivors of a cardiac arrest frequently develop severe postanoxic encephalopathy. Derangements in cerebral blood after return of spontaneous circulation play an important role in the pathogenesis of postanoxic encephalopathy. In the present study we examine the effect of mild therapeutic hypothermia on cerebral blood flow and carbondioxide reactivity in patients after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* GCS after return of circulation < 7
* Induced mild hypothermia for 24 hours
* primary rhythm ventricular fibrillation

Exclusion Criteria:

* Thrombolysis
* Cardiogenic shock with expected survival < 24 hrs
* Pregnancy
* No informed consent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after cardiac arrest, comatose and treated with therapeutic hypothermia
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Hoedemaekers, MD PhD, Principal Investigator — Radboud University Medical Center; Johannes van der Hoeven, MD PhD, Study Director — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands